CLINICAL TRIAL: NCT05225805
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Assess the Safety and Pharmacokinetics Following Single Doses of Oral and Intravenous Xenleta (Lefamulin) in Adult Patients With Cystic Fibrosis
Brief Title: Study to Assess the Safety and PK of Oral and IV Xenleta in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NAB-BC-3781-1014
Record Dates: First submitted 2022-01-07; First posted 2022-02-07 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lefamulin

STUDY DESIGN:
Intervention Model Description: Open-label, Crossover Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive one dose of 150 mg lefamulin IV followed by one dose of 600 mg lefamulin oral
  Interventions: Drug: Lefamulin
- Group B (Experimental): Group B will receive one dose of 600 mg lefamulin oral followed by one dose of 150 mg lefamulin IV
  Interventions: Drug: Lefamulin

INTERVENTIONS:
Drug: Lefamulin — Antibiotic
  Other Names: BC-3781

SUMMARY:
This study is intended to assess the pharmacokinetic (PK) and safety of a single dose of IV and oral formulations of lefamulin in adults with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Staphylococcus aureus is one of the most common causative pathogens associated with exacerbations of CF. Current treatment guidelines for the management of exacerbations of CF caused by S. aureus recommend the use of unapproved antibacterial agents. Further, many of the recommended treatments can only be administered via the IV route and/or have limitations due to safety and tolerability. Lefamulin is a novel, first-in-class, IV and oral pleuromutilin antimicrobial agent that has been demonstrated to be highly potent against S. aureus, including Methicillin-resistant Staphylococcus aureus (MRSA) and strains obtained from patients with CF. Cystic fibrosis patients have altered drug distribution and elimination kinetics for many antimicrobials relative to patients without CF. While the advent of Cystic fibrosis transmembrane conductance regulator (protein) (CFTR) modulators has resulted in improved lung function and had a positive impact on the quality of life of CF patients, limited data have been published describing the impact of the concomitant use of CFTR modulators and commonly used antibacterial agents.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Adult patients, ≥ 18 years of age.
3. Genetic confirmation of CF diagnosis by a report from a genetic test, such as "F508 deletion detected."
4. Weight > 40 kgs.
5. Forced expiration volume (FEV)1 > 40% predicted, as measured during the most recent evaluation.
6. Mentally and physically able to participate in the study as determined by the Investigator, ie, clinically stable with no significant changes in health status within 28 days prior to, and including, Day 1.
7. Vital signs within the following ranges:

   1. Tympanic temperature, < 38°C
   2. Systolic blood pressure, 90 to 160 mmHg
   3. Diastolic blood pressure, 50 to 90 mmHg
   4. Heart rate < 100 beats per minute at rest
   5. Respiration rate 12 to 20 breaths per minute
   6. Oxygen saturation to be documented. No selection criteria; supplemental oxygen use is acceptable.
8. Negative beta-human chorionic gonadotropin (β-hCG) urine or serum pregnancy test for females of childbearing potential.
9. Willing to commit to acceptable methods of contraception as defined in the protocol.

Exclusion Criteria:

1. Known history of chronic liver or biliary disease, Gilbert's syndrome, or any of the following at Screening: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN), total bilirubin > 1.5 x ULN.
2. Prolonged baseline corrected QT interval corrected according to Fridericia (QTcF) defined as > 440 ms (females) and > 430 ms (males).
3. Family history or presence of prolonged QTc syndrome, Torsades de Pointes, or known conduction defects (eg, bundle branch block, atrioventricular block).
4. Use of Orkambi® (lumacaftor/ivacaftor) within 28 days prior to Day 1.
5. Use of cytochrome P450 (CYP)3A substrates that prolong the QT interval within 24 hours prior to Day 1.
6. Use of strong and moderate Cytochrome P450 (CYP3A) inducers or P-glycoprotein (P-gp) inducers within 28 days prior to Day 1.
7. Use of strong inhibitors of CYP3A4 within 24 hours prior to Day 1.
8. Serum potassium level below the normal reference range at Screening.
9. Known allergy to pleuromutilin class of antibiotic or any of the excipients of the lefamulin formulations.
10. Consumption of grapefruit, grapefruit juice, grapefruit products, pomelo, or Seville oranges within 24 hours before Day 1.
11. Use of vaporized nicotine or cannabidiol products, smoking (regularly or intermittently) more than 5 cigarettes (or equivalent) per day, or any use of tobacco other than in cigarettes or cigars within 28 days of Day 1.
12. Positive blood test for hepatitis C, human immunodeficiency virus (HIV), or hepatitis B antigen or core antibody (indicating active infection).
13. Positive test for drugs of abuse or alcohol at Screening or Day 1 that cannot be satisfactorily supported by medical history.
14. Use of an investigational product within the 30 days prior to Day 1 (3 months prior to Day 1 if the study drug was a new chemical entity).
15. Difficulty swallowing tablets.
16. Females who are pregnant or breastfeeding.
17. Does not have suitable venous access for multiple venipuncture or cannulation.
18. Any medical, psychological, cognitive, social, or legal conditions that, in the opinion of the Investigator, would interfere with the patient's ability to give an informed consent and/or participate fully in the study.
19. Any other reason, in the opinion of the Investigator, the patient is unsuitable to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Kansas School of Medicine, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - New York Medical College, Valhalla, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State University College of Medicine, Hershey, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sawicki GS, Wicha WW, Hiley TS, Close NC, Gelone SP, Guico-Pabia CJ. Safety and Pharmacokinetics Following Oral or Intravenous Lefamulin in Adults With Cystic Fibrosis. Clin Ther. 2024 Feb;46(2):96-103. doi: 10.1016/j.clinthera.2023.12.002. Epub 2024 Jan 8. PMID 38195348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple investigative sites in United States.
Pre-assignment Details: A total of 13 subjects (4 females, 9 males) was enrolled in the study and treated in the study NAB-BC-3781-1014. One subject failed screening.
Groups:
- Group A (IV-Oral): Group A will receive single dose of lefamulin 150 mg IV infusion in 250 mL citrate buffered saline over 1 hour followed by lefamulin 600-mg immediate-release (IR) tablet orally in the fasted state.
  Lefamulin: Antibiotic
- Group B (Oral-IV): Group B will receive single dose of lefamulin 600 mg immediate-release (IR) tablet orally in the fasted state followed by single dose of lefamulin 150 mg IV infusion in 250 mL citrate buffered saline over 1 hour.
  Lefamulin: Antibiotic
Period: Overall Study
Arm/Group | Group A (IV-Oral) | Group B (Oral-IV)
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All 13 adult subjects received at least 1 dose of IMP and were included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (IV-Oral) | Group B (Oral-IV) | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.0 (11.14) | 31.1 (9.01) | 29.2 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Median for Lefamulin and Its Main Metabolite BC-8041 for PK Plasma Parameter Tmax in Cystic Fibrosis (CF) Patients.
Description: Appropriate non-compartmental techniques were used to obtain estimates for the PK parameter Tmax in plasma for lefamulin and its metabolite BC-8041.
  Time to reach maximum plasma concentration of lefamulin following drug administration (Tmax)
  Tmax will be determined by direct inspection of the concentration versus time data by WinNonlin.
Time Frame: Pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 2 hrs, 4 hrs, 8 hrs, 12 hrs & 24 hrs Post-dose
Population: Pharmacokinetic (PK) Population: All 13 adult subjects completed both periods of the study. Plasma samples from 13 subjects were analyzed for lefamulin and BC-8041.
Measure: Median (Full Range); unit: hours
Groups:
- Lefamulin Oral Treatment: Lefamulin as a 600-mg IR tablet. The oral treatment will be swallowed whole with 6 to 8 ounces of water at least 1 hour before or 2 hours after a meal.
- Lefamulin IV Treatment: Lefamulin 150 mg in 250 mL citrate buffered saline IV infusion over 1 hour.
Arm/Group | Lefamulin Oral Treatment | Lefamulin IV Treatment
Number analyzed (Participants) | 13 | 13
hours
  Lefamulin | 2.00 [0.983 to 3.900] | 0.583 [0.500 to 1.717]
  Lefamulin metabolite BC-8041 | 1.517 [1.017 to 4.017] | 1.500 [0.933 to 1.817]

2. Primary Outcome: The Key Geometric Mean for Lefamulin and Its Main Metabolite BC-8041 for PK Plasma Parameter Cmax in CF Patients.
Description: Appropriate non-compartmental techniques will be used to obtain estimates for the PK parameter Cmax in plasma for lefamulin and its metabolite BC-8041.
  Maximum observed plasma concentration (Cmax)
  Cmax was determined by direct inspection of the concentration versus time data by WinNonlin.
Time Frame: Pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 2 hrs, 4 hrs, 8 hrs, 12 hrs & 24 hrs Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Lefamulin Oral Treatment | Lefamulin IV Treatment
Number analyzed (Participants) | 13 | 13
mg/L
  Lefamulin | 1.314 (0.308) | 1.924 (0.417)
  Lefamulin Metabolite BC-8041 | 0.351 (0.417) | 0.030 (0.470)

3. Primary Outcome: The Key Geometric Mean for Lefamulin and Its Main Metabolite BC-8041 for PK Plasma Parameter AUC(0-last) in CF Patients.
Description: Appropriate non-compartmental techniques will be used to obtain estimates for the PK parameter (AUC0-last) in plasma for lefamulin and its metabolite BC-8041.
  AUC calculations will be performed using the linear/log trapezoidal rule. AUC0-last will be calculated between t0hr and the last measurable concentration.
  Area under the drug concentration curve from time zero (0 h) to 24 h (AUC0-last)
Time Frame: Pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 2 hrs, 4 hrs, 8 hrs, 12 hrs & 24 hrs Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg·h/L
Groups:
- Oral Treatment: Lefamulin as a 600-mg IR tablet. The oral treatment will be swallowed whole with 6 to 8 ounces of water at least 1 hour before or 2 hours after a meal.
- IV Treatment: Lefamulin 150 mg in 250 mL citrate buffered saline IV infusion over 1 hour.
Arm/Group | Oral Treatment | IV Treatment
Number analyzed (Participants) | 13 | 13
mg·h/L
  Lefamulin | 6.881 (0.380) | 6.220 (0.286)
  Lefamulin Metabolite BC-8041 | 1.990 (0.442) | 0.232 (0.536)

4. Primary Outcome: The Key Geometric Mean for Lefamulin and Its Main Metabolite BC-8041 for PK Plasma Parameter AUC(0-inf) in CF Patients.
Description: Appropriate non-compartmental techniques will be used to obtain estimates for PK parameter AUC(0-inf) in plasma for lefamulin and its metabolite BC-8041.
  AUC calculations will be performed using the linear/log trapezoidal rule. AUC(0-inf) will be will be calculated between t0hr and infinity.
  Area under the drug concentration curve from time zero (0 h) to infinity (AUC(0-inf)
Time Frame: Pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 2 hrs, 4 hrs, 8 hrs, 12 hrs & 24 hrs Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg·h/L
Arm/Group | Lefamulin Oral Treatment | Lefamulin IV Treatment
Number analyzed (Participants) | 13 | 13
mg·h/L
  Lefamulin | 7.277 (0.384) | 6.568 (0.286)
  Metabolite BC-8041 | 2.095 (0.448) | 0.272 (0.517)

5. Primary Outcome: The Key Geometric Mean for Lefamulin and Its Main Metabolite BC-8041 for PK Plasma Parameter t1/2 in CF Patients.
Description: Appropriate non-compartmental techniques will be used to obtain estimates for thr PK parameter t1/2 in plasma for lefamulin and its metabolite BC-8041.
  Apparent elimination half-life calculated as ln(2)/ke (t½)
Time Frame: Pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 2 hrs, 4 hrs, 8 hrs, 12 hrs & 24 hrs Post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oral Treatment | IV Treatment
Number analyzed (Participants) | 13 | 13
hours
  Lefamulin | 6.422 (0.182) | 6.297 (0.188)
  Metabolite BC-8041 | 5.796 (0.175) | 8.128 (0.176)

ADVERSE EVENTS:
Time Frame: Up-to Follow-up (4 to 7 days after the final dose).
Description: Safety analysis set (SfAS): All subjects who receive any full or partial dose of lefamulin. The SfAS will be used for the analysis of safety data.
Groups:
- Total: Lefamulin oral treatment + Lefamulin IV treatment
  Lefamulin as a 600-mg IR tablet. The oral treatment will be swallowed whole with 6 to 8 ounces of water at least 1 hour before or 2 hours after a meal.
  Lefamulin 150 mg in 250 mL citrate buffered saline IV infusion over 1 hour.
Arm/Group | Lefamulin Oral Treatment | Lefamulin IV Treatment | Total
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 4/13 | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lefamulin Oral Treatment (N=13) | Lefamulin IV Treatment (N=13) | Total (N=13)
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Infusion site erythema (General disorders) | 0 | 1 | 1
Infusion site pain (General disorders) | 0 | 1 | 1
Cystic fibrosis gastrointestinal disease (Congenital, familial and genetic disorders) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT05225805/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT05225805/SAP_001.pdf